CLINICAL TRIAL: NCT05723458
Title: The Joint Effects of Turmeric, Black Seeds, Flaxseed and Medicago Sativa for Relieving Symptoms of Knee Osteoarthritis: A Phase 1-2 Randomized, Double-Blind, Placebo-Controlled Clinical Trial
Brief Title: Turmeric, Black Seeds, Flaxseed and Medicago Sativa in Knee Osteoarthritis
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tabriz University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Dr. Saeid Safiri, Principal Investigator, Tabriz University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 70180
Record Dates: First submitted 2023-01-17; First posted 2023-02-10 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Knee Osteoarthritis
Keywords: Knee osteoarthritis; Turmeric; Black Seeds; Flaxseed; Medicago Sativa
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cream containing Turmeric, Black Seeds, Flaxseed, and Medicago Sativa (Active Comparator)
  Interventions: Combination Product: Cream
- Placebo cream containing vaseline (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Combination Product: Cream — A cream containing Turmeric, Black Seeds, Flaxseed, and Medicago Sativa
  Arms: Cream containing Turmeric, Black Seeds, Flaxseed, and Medicago Sativa
Drug: Placebo — Placebo cream containing vaseline
  Arms: Placebo cream containing vaseline

SUMMARY:
This study investigates the safety and combined effect of Turmeric, Black Seeds, Flaxseed, and Medicago Sativa for relieving symptoms of knee osteoarthritis compared to the placebo group.

DETAILED DESCRIPTION:
The present double-blind, randomized and placebo-controlled study will be conducted on patients with knee osteoarthritis to evaluate the safety and efficacy of a combined cream of Turmeric, Black Seeds, Flaxseed, and Medicago Sativa for relieving symptoms of knee osteoarthritis. The primary endpoints will be the pain, stiffness, and physical function subscales of the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) criteria, subject global evaluation (SGE), and the overall WOMAC score. Also, the secondary endpoints of this study include an evaluation of the quality of life, quality of sleep, and Functional Capacity Classification.

A pilot study with 30 participants per arm will be conducted to estimate the final sample size. Adults over 40 years of age who have had OA for at least 6 months, and whose OA diagnosis meets the American College of Rheumatology criteria will be eligible to participate in the present study. Participants will be randomized in the intervention or placebo group to use a cream containing 95% vaseline and 5% mixed extract of Turmeric, Black Seeds, Flaxseed, and Medicago Sativa as intervention or cream of vaseline solely as a placebo. The cream will be administrated topically three times daily (9 AM, 3 PM, and 9 PM) for up to 12 weeks. The efficacy and safety of the creams will be measured during visits on days 30, 60, and 90 (final visit). Also, the complications and adherence of patients to intervention will be checked on days 15, 45, and 75 by telephonic discussion. The analysis will be performed based on the intent-to-treat method.

ELIGIBILITY:
Inclusion Criteria:

* At least 6 months of diagnosis of knee osteoarthritis, and whose OA diagnosis meets the American College of Rheumatology criteria,
* Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) pain subscale baseline value of ≥ 9 (0-20 scale),
* Functional Capacity Classification of I-III,
* Radiograph evidence of OA in the target knee with a Kellgren-Lawrence score of 2 or 3,
* Morning stiffness of <30 min duration or crepitus on active motion, which are present upon examination.

Exclusion Criteria:

* Evidence of other conditions or diseases of the skin or joints,
* Evidence of partial or complete knee joint replacement or anticipated joint replacement in the target knee,
* Contraindications to the use of non-steroidal anti-inflammatory drugs (NSAIDs) or who use anticoagulant therapy that prohibits them from using NSAIDs,
* Pregnancy, planning to become pregnant or breastfeeding during the study period,
* Ischemic heart disease, heart failure, end-stage cirrhosis, end-stage renal failure, or psychiatric conditions that prevent an adequate evaluation of the study outcomes,
* Insufficient cognitive functioning to participate and complete the questionnaires,
* Unable or unwilling to follow up and complete the study pathway,
* Having active cancer undergoing treatment that prevents the evaluation of the outcome measures,
* A history or diagnosis of other arthritic conditions, such as rheumatoid arthritis, joint and bone deformities, fibromyalgia, and/or other inflammatory and immune system disorders,
* Type I or II diabetes or obesity (body mass index ≥ 39),
* Suffering from painful conditions or frequent headaches requiring the use of systemic opiates or derivatives, or the need for additional NSAID or COX-2 inhibitors,
* Receiving systemic or intra-articular corticosteroid injections.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Pain subscale of the Western Ontario and McMaster Universities Osteoarthritis criteria | Day 0, 30, 60, 90 post intervention
  Change in pain subscale of the Western Ontario and McMaster Universities Osteoarthritis criteria in response to intervention. The pain subscale scores range from 0 (no pain with all 5 activities, ie, flat surface walking, stairclimbing, at night, sitting or lying, standing) to 20 (extreme pain with all 5 activities). Higher scores represent worse situation.
Stiffness subscale of the Western Ontario and McMaster Universities Osteoarthritis criteria | Day 0, 30, 60, 90 post intervention
  Change in stiffness subscale of the Western Ontario and McMaster Universities Osteoarthritis criteria in response to intervention. The scores for stiffness subscale range from 0 to 8 and higher scores represent worse situation.
Physical function subscale of the Western Ontario and McMaster Universities Osteoarthritis criteria | Day 0, 30, 60, 90 post intervention
  Change in physical function subscale of the Western Ontario and McMaster Universities Osteoarthritis criteria in response to intervention. The scores for physical function subscale range from 0 to 68 and higher scores represent more physical limitation.
Overall Western Ontario and McMaster Universities Osteoarthritis score | Day 0, 30, 60, 90 post intervention
  Change in overall Western Ontario and McMaster Universities Osteoarthritis score in response to intervention. The scores for each subscale are summed up, with a possible score range of 0-96 and higher scores indicate worse pain, stiffness, and functional limitations.
Subjective Global Evaluation | Day 0, 30, 60, 90 post intervention
  Change in Subjective Global Evaluation in response to intervention. According to the Subjective Global Evaluation questionnaire, the status of the patients is determined as normal (0), mild (1+), moderate (2+) or severe (3+) malnutrition.

SECONDARY OUTCOMES:
Quality of life index | Day 0, 30, 60, 90 post intervention
  Change in quality of life index in response to intervention
Pittsburgh Sleep Quality Index score | Day 0, 30, 60, 90 post intervention
  Change in the Pittsburgh Sleep Quality Index score in response to intervention. The sleep component scores are summed to yield a total score ranging from 0 to 21 with the higher total score indicating worse sleep quality.
Functional Capacity Classification | Day 0, 30, 60, 90 post intervention
  Change in Functional Capacity Classification in response to intervention. It is measured in a 4 point Likert scale and higher values represent worse situation.

CONTACTS AND LOCATIONS:
Locations (1):
- Imam Reza hospital and clinic of Salamat, Tabriz, AzarbayejaneShargi, Iran

IPD SHARING:
Plan to Share IPD: No